CLINICAL TRIAL: NCT00256594
Title: Evaluation of an Outpatient Modified Paper Prescription Form in 4 Rural States to Address the Public Health Problem of Prescribing Error
Brief Title: Evaluation of an Outpatient Modified Prescription Form
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Kennedy, Assistant Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1 R04RH05814-01-00
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Medication Errors
Keywords: Medical Errors; Medication Errors; Prescriptions, Drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: prescription form — Two prescription pads contained modified forms and two prescription pads were similar to the prescription pads the prescriber had been using. Providers completed 100 standard and 100 modified prescriptions

SUMMARY:
The purpose of this study is to determine if a modified paper prescribing form decreases prescribing errors compared to a traditional or standard paper prescribing form.

DETAILED DESCRIPTION:
The broad goal of this proposal is to reduce outpatient prescribing errors in rural primary care practices. Although computerized technology is available for prescribing, it has not yet been implemented in most settings. Additionally, rural prescribers will likely be the last to have the means to adopt this technology. Due to the substantial morbidity and mortality in the United States caused by outpatient medication errors, there is an urgent need for low-cost solutions. This research plan will evaluate a modified paper prescription form that may be implemented in rural primary care settings cheaply and quickly with the goal of outpatient prescription error reduction.

The specific aims of this project are:

1. To determine if a modified paper prescription form decreases overall prescribing errors compared to a standard paper prescription form
2. To determine if a modified paper prescription form decreases omission errors compared to a standard paper prescription form
3. To determine prescriber satisfaction with the modified prescription form

Rural prescribers from four states will be randomly recruited to write prescriptions on standard and modified forms. Prescription duplicates of both types will be analyzed for errors. Prescriber satisfaction with the modified form will be evaluated using surveys and focus groups.

Medication errors are a public health problem. Low-cost technology that is shown to reduce medication errors would benefit all rural patients who receive prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Must be a physician, nurse practitioner, or physician assistant with a current license to write outpatient prescriptions
* Must practice in Family Practice, Internal Medicine, or Pediatrics
* Must practice in rural Vermont, West Virginia, South Dakota, or Montana
* Must write outpatient paper prescriptions
* Must write prescriptions in English

Exclusion Criteria:

* Not licensed to write prescriptions
* Practice in a specialty, inpatient, or long term care setting
* Do not write paper prescriptions
* Do not write prescriptions in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-08; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
error rates of standard versus modified prescriptions per prescriber | 200 prescriptions each

CONTACTS AND LOCATIONS:
Overall Officials: Amanda G Kennedy, PharmD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Division of General Internal Medicine, Burlington, Vermont, United States

REFERENCES:
- [Background] Kennedy AG, Littenberg B. A modified outpatient prescription form to reduce prescription errors. Jt Comm J Qual Saf. 2004 Sep;30(9):480-7. doi: 10.1016/s1549-3741(04)30056-0. PMID 15469125
- [Result] Kennedy AG, Littenberg B, Callas PW, Carney JK. Evaluation of a modified prescription form to address prescribing errors. Am J Health Syst Pharm. 2011 Jan 15;68(2):151-7. doi: 10.2146/ajhp100063. PMID 21200063
- [Result] Kennedy AG, Senders JW, Sellen K, Littenberg B, Callas PW, Carney JK. Perception of drug-name legibility by pharmacists and pharmacy technicians. Am J Health Syst Pharm. 2009 May 1;66(9):794-5. doi: 10.2146/ajhp080189. No abstract available. PMID 19386937